CLINICAL TRIAL: NCT04669782
Title: Osteocalcin in Bone Metabolism and Aging: Effect of Vitamin K Supplementation on Circulating Levels of Osteocalcin, on Glucose and Energy Metabolism and on Muscle Mass and Function
Brief Title: Effect of Vitamin K Supplementation on Circulating Levels of Osteocalcin on the Bone Metabolism and Aging
Acronym: OstMARK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistics/management problems at the recruiting center
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OstMARK
Record Dates: First submitted 2020-11-24; First posted 2020-12-17 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Bone Metabolism Disorder; Aging Disorder; Osteoporosis
Keywords: osteocalcin; vitamin k
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Vitamin K; Teriparatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with osteoporosis treated with teriparatide + Vitamin K (Experimental): Patients will have to take teriparatide (standard of care) + Vitamin K (MK7) at the dosage of 375 microg / day
  Interventions: Dietary Supplement: Vitamin K (MK7); Drug: Teriparatide
- Patients with osteoporosis treated with teriparatide (Active Comparator): Patients will have to take teriparatide (standard of care)
  Interventions: Drug: Teriparatide
- Controls (No Intervention): Subject without osteoporosis, no treatment will be administered.

INTERVENTIONS:
Dietary Supplement: Vitamin K (MK7) — MK-7 will be administered at a dose of 375 microg / day
  Arms: Patients with osteoporosis treated with teriparatide + Vitamin K
Drug: Teriparatide — Teriparatide will be administered as standard of care
  Arms: Patients with osteoporosis treated with teriparatide; Patients with osteoporosis treated with teriparatide + Vitamin K

SUMMARY:
This is an interventional study on nutraceuticals. It is a randomized controlled, open-label, prospective, single-center study that involves the enrollment of 82 patients with osteoporosis and 41 subjects without osteoporosis.

The hypothesis the decarboxylated form of Osteocalcin (OC), called GluOC, represents a clinically useful marker for monitoring the effects of supplementation with vitamin K in association with anabolic treatment with teriparatide will be analyzed not only on bone but also on skeletal muscle and energy metabolism in patients with severe osteoporosis.

DETAILED DESCRIPTION:
Background:

OC, also known as bone-Gla-protein (BGP), is the main non-collagen protein of the extracellular matrix in mineralized tissues. It is synthesized by osteoblasts, odontoblasts, and hypertrophic chondrocytes and, through its negative charges, binds calcium and regulates the formation of hydroxyapatite crystals.

In humans, circulating OC levels negatively correlate with fasting blood glucose and insulin, Homeostatic Model Assessment for Insulin Resistance (HOMA-IR), body mass index (BMI), hyperlipidemia, and circulating concentrations of leptin. Weight loss (resulting from diet and / or physical activity) improves metabolic profile and muscle strength and increases OC levels.

It's interesting to note that high plasma levels of vitamin K or dietary supplementation (MK-7, the natural derivative of vitamin K2), correlate with a reduction in the loss of bone mass and quality. In addition, short-term (1 week) and long-term (3 years) vitamin K supplementation improves insulin resistance in both young and old males and high vitamin K consumption is associated with reduced insulin resistance and reduced risk of developing type 2 mellitus diabetes.

Recently, it has been reported in mice that the combination of teriparatide (TPT) and vitamin K is more effective than ionotherapy in improving bone formation, bone density and strength, and in inhibiting bone resorption.

Given the putative relevance of the decarboxylated form of OC, GluOC, in the endocrine interaction between bone and organs responsible for the management of energy resources (e.g. endocrine pancreas, skeletal muscle and adipose tissue) whose function is deregulated in elderly subjects and in the syndrome of fragility, this study aims to define a role of supplementation with vitamin K in osteoporosis, another condition characterizing the frailty of the elderly, on the endocrine function of bone tissue and the consequent effects on energy metabolism.

There is various evidence regarding the usefulness of using the decarboxylated form of OC as a biomarker for monitoring the response to anti-osteoporotic treatments. In particular, the circulating levels of GluOC respond both to osteometabolic treatments (teriparatide) and to supplementation with vitamin K, in a more relevant way than to total osteocalcin.

Study design and treatment:

The study includes the following phases:

1. enrollment of controls, after obtaining informed consent.
2. enrollment of patients, after obtaining informed consent.
3. randomization for the patient group
4. prescription teriparatide +/- Vitamin K depending on the group to which it belongs
5. re-evaluation of patients after 6, 12 and 18 months of treatment

The group of patients randomized to the teriparatide + Vitamin K / Menaquinone MK-7 arm will have to take MK-7 at a dose of 375 microg / day.

Randomization:

Patients with osteoporosis will be randomized 1: 1 to one of two treatment groups:

* Teriparatide + Vitamin K
* Teriparatide

The randomization list will be generated with SAS 9.4 software (SAS Institute Inc., Cary, USA) and foresees the presence of blocks.

Statistical Analysis:

The analysis of the covariance will be performed to evaluate the effect of treatment with and without vitamin K / MK-7 on the primary endpoint measured at 18 months, adjusting for its baseline value (α = 0.05, two-tailed test). The results will also be described in terms of means and 95% confidence intervals both of the absolute values of GluOC at 18 months and of its variations from baseline. This approach will also be followed for the evaluation of the effect of the intake of vitamin K / MK-7 on the secondary endpoints defined by the OC isoforms.

The association between GluOC and Gla-type Osteocalcin (GlaOC) levels at 18 months (and changes from baseline) with respect to the markers of energy, bone and muscle metabolism measured at 18 months will also be explored through a linear regression model.

ELIGIBILITY:
Inclusion Criteria

Inclusion criteria for the group "Patients with osteoporosis":

* Age ≥ 65 years
* Serum levels of 25OHD> 30 ng / ml (as per clinical practice)
* Adequate calcium intake (assessed by questionnaire)
* Diagnosis of severe primary osteoporosis
* Criteria for the prescription and reimbursement of treatment with Teriparatide 20 microg / day subcutaneous according to the Italian Agency of Pharma (AIFA) 79
* Patient suitable for treatment with MK-7
* Informed consent freely acquired before the person was enrolled

Inclusion criteria for the group "subjects without osteoporosis":

* Age ≥ 65 years
* Serum levels of 25OHD> 30 ng / ml (as per clinical practice)
* Adequate calcium intake (assessed by questionnaire).
* Informed consent freely acquired before the person was enrolled

Exclusion Criteria:

Exclusion criteria for the group of "Patients with osteoporosis":

* causes of secondary osteoporosis: current glucocorticoid therapy, active and uncontrolled rheumatic diseases, endogenous hypercortisolism, uncontrolled hyperthyroidism or hypothyroidism (except known hypothyroidism well compensated with L-thyroxine), chronic renal failure (IRC) with glomerular filtration rate (GFR) <30 ml / min, multiple myeloma, liver failure (chronic liver disease of CHILD class B and C), heart failure (New York Heart Association, also said NHYA) NHYA> 2, active neoplasms, type 1 and type 2 diabetes mellitus
* ongoing therapies: glucocorticoids, antiepileptics, aromatase inhibitors and similar gonadotropin-releasing hormone (GnRH, contraindicated for teriparatide).

Exclusion criteria for the group "subjects without osteoporosis":

* ongoing therapies: glucocorticoids, antiepileptics, diphosphonates, teriparatide, denosumab, statins, oral or injective hypoglycemic agents, aromatase inhibitors, similar GnRH or other oncological therapies
* diagnosis of osteoporosis (according to World Health Organization, WHO) T-score <-2.5 standard deviation (SD), at any site evaluated with ''Dual-Energy X-ray Absorptiometry'' (DXA)
* diagnosis of sarcopenia (according to ''Appendicular Skeletal Muscle Mass'', ASMMI) ASMMI <7.59 kg / m2 for males and 5.47 kg / m2 for females evaluated with DXA
* diagnosis of IRC with estimated GFR <30 ml / minute, liver failure (chronic liver disease of CHILD class B and C), heart failure with NHYA> 2 , active neoplasms, endocrinopathies (except known hypothyroidism well compensated with L-thyroxine ), type 1 and type 2 diabetes mellitus.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 99 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2024-07-04 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Circulating levels of GluOC | 18 months
  Circulating levels of GluOC measured after 18 months of treatment with vitamin K

SECONDARY OUTCOMES:
Circulating levels of OC isoforms | 18 months
  Circulating levels of OC isoforms measured after 18 months of treatment with vitamin K

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Galeazzi IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Airoldi C, Giovannardi S, La Ferla B, Jimenez-Barbero J, Nicotra F. Saturation transfer difference NMR experiments of membrane proteins in living cells under HR-MAS conditions: the interaction of the SGLT1 co-transporter with its ligands. Chemistry. 2011 Nov 25;17(48):13395-9. doi: 10.1002/chem.201102181. Epub 2011 Oct 27. No abstract available. PMID 22031470
- [Background] Anastasilakis A, Goulis DG, Koukoulis G, Kita M, Slavakis A, Avramidis A. Acute and chronic effect of teriparatide on glucose metabolism in women with established osteoporosis. Exp Clin Endocrinol Diabetes. 2007 Feb;115(2):108-11. doi: 10.1055/s-2007-967090. PMID 17318770
- [Background] Ebina K, Hashimoto J, Shi K, Kashii M, Hirao M, Yoshikawa H. Comparison of the effect of 18-month daily teriparatide administration on patients with rheumatoid arthritis and postmenopausal osteoporosis patients. Osteoporos Int. 2014 Dec;25(12):2755-65. doi: 10.1007/s00198-014-2819-x. Epub 2014 Aug 1. PMID 25082556
- [Background] Ferron M, McKee MD, Levine RL, Ducy P, Karsenty G. Intermittent injections of osteocalcin improve glucose metabolism and prevent type 2 diabetes in mice. Bone. 2012 Feb;50(2):568-75. doi: 10.1016/j.bone.2011.04.017. Epub 2011 Apr 29. PMID 21550430
- [Background] Grasso D, Corsetti R, Lanteri P, Di Bernardo C, Colombini A, Graziani R, Banfi G, Lombardi G. Bone-muscle unit activity, salivary steroid hormones profile, and physical effort over a 3-week stage race. Scand J Med Sci Sports. 2015 Feb;25(1):70-80. doi: 10.1111/sms.12147. Epub 2013 Oct 31. PMID 24433517
- [Background] Gundberg CM, Lian JB, Booth SL. Vitamin K-dependent carboxylation of osteocalcin: friend or foe? Adv Nutr. 2012 Mar 1;3(2):149-57. doi: 10.3945/an.112.001834. PMID 22516722
- [Background] Knapen MHJ, Jardon KM, Vermeer C. Vitamin K-induced effects on body fat and weight: results from a 3-year vitamin K2 intervention study. Eur J Clin Nutr. 2018 Jan;72(1):136-141. doi: 10.1038/ejcn.2017.146. Epub 2017 Sep 27. PMID 28952607